CLINICAL TRIAL: NCT00886275
Title: Comparing the Effect of Dexmedetomidine With Midazolam on Sedation, Oxidative Stress, and Microcirculation in Intensive Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200901037M
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Sedation; Oxidative Stress
Keywords: Postoperative sedation in intensive care
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam
- Dexmedetomidine, Midazolam (Experimental): Combination
  Interventions: Drug: Dexmedetomidine, Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — The loading dose of dexmedetomidine is 0.5 mcg/kg over 10 minutes as needed. Then, continuous infusion of 0.2-0.7 mcg/kg/h dexmedetomidine is used to maintain RASS between 0 to -3.
  Arms: Dexmedetomidine
Drug: Midazolam — The loading dose of midazolam is 0.05 mg/kg over 10 minutes as needed. Then, continuous infusion of 20-300 mcg/kg/h midazolam is used to maintain RASS between 0 to -3.
  Arms: Midazolam
Drug: Dexmedetomidine, Midazolam — The loading doses are dexmedetomidine 0.25 mcg/kg and 0.025 mg/kg of midazolam over 10 minutes. Then, continuous infusion of 0.1-0.7 mcg/kg/h dexmedetomidine and 10-300 mcg/kg/h midazolam is used to maintain RASS between 0 to -3.
  Arms: Dexmedetomidine, Midazolam

SUMMARY:
In intensive care unit, patients suffered pain and anxiety from mechanical ventilation, presence of endotracheal tube, central venous catheter, postoperative wound, and invasive procedures. Adequate analgesia and sedation can reduce pain and anxiety. However, traditional sedatives carry the risk of unstable hemodynamic status, respiratory depression, increased mechanical ventilation time, incidence of delirium, and length of ICU stay. Dexmedetomidine is a highly selec¬tive α2-adrenergic receptor agonist which causes sedative effects and reduces opioid requirements in the perioperative period. Memis et al had found that dexmedetomidine may prevent inflammatory effects in sepsis patients during sedation. Oxidative stress status is related to the inflammatory response. Moreover, oxidative stress may result in dysfunction of microcirculation. Dysfunction of microcirculation may cause vasoconstriction or microthrombosis, and it will impair tissue perfusion and result in organ dysfunction. The goal of this study is to compare the effects of dexmedetomidine and midazolam on requirement of analgesics, weaning parameter, hemodynamic status, time of extubation, incidence of delirium, and length of ICU stay, oxidative stress status, and microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is older than 18 years old and less than 80 years old
* Patient who is admitted to intensive care unit with artery line
* Patient's hemodynamic status is stable under adequate management and absence of signs of shock
* Patient who has understood the inform consent and agree to participate this study

Exclusion Criteria:

* Patient's hemodynamic status is unstable in spite of adequate management or presence of signs of shock
* Patient who has a past history of allergy to study drugs
* Patient who has renal failure or requires renal replacement therapy
* Patient who has liver cirrhosis or liver failure
* Patient who has participated in any other investigational study of other drugs currently
* Female patient who is pregnant or considers breast feeding currently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time to extubation | hour

SECONDARY OUTCOMES:
ICU Stay Weaning parameter | Hour

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan